CLINICAL TRIAL: NCT01939028
Title: Sentinel Lymph Node Mapping for Endometrial Cancer
Brief Title: Lymph Node Mapping in Patients With Newly Diagnosed Endometrial Cancer Undergoing Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE9813; NCI-2013-01309 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-07-10; First posted 2013-09-11 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Stage I Endometrial Carcinoma; Stage II Endometrial Carcinoma; Stage III Endometrial Carcinoma; Stage IV Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Sentinel Lymph Node Biopsy; iso-sulfan blue; Indocyanine Green; Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (SLN mapping, biopsy, surgery) (Experimental): Patients undergo SLN mapping using isosulfan blue and/or indocyanine green solution injected directly into the cervix. Following SLN identification and biopsy, patients undergo hysterectomy, bilateral salpingo-oophorectomy, and/or complete pelvic lymphadenectomy. Patients expressing SLN positive for metastasis undergo para-aortic lymphadenectomy.
  Interventions: Procedure: lymph node mapping; Procedure: sentinel lymph node biopsy; Drug: isosulfan blue; Drug: indocyanine green solution; Procedure: therapeutic conventional surgery; Procedure: lymphadenectomy

INTERVENTIONS:
Procedure: lymph node mapping — Undergo lymph node mapping using isosulfan blue and/or indocyanine green solution
Procedure: sentinel lymph node biopsy — Undergo SLN biopsy
  Other Names: sentinel node biopsy
Drug: isosulfan blue — Undergo lymph node mapping using isosulfan blue and/or indocyanine green solution
  Other Names: Lymphazurin; N-[4-[4-(diethylamino)phenyl] (2,5-disulfophenyl) Methylene]-2,5-cyclohexadien-1-ylidene]-N-ethylethanaminium hydroxide
Drug: indocyanine green solution — Undergo lymph node mapping using isosulfan blue and/or indocyanine green solution
  Other Names: IC-GREEN; ICG solution
Procedure: therapeutic conventional surgery — Undergo hysterectomy, bilateral salpingo-oophorectomy and/or complete pelvic lymphadenectomy
Procedure: lymphadenectomy — Undergo para-aortic lymphadenectomy

SUMMARY:
This clinical trial studies lymph node mapping in patients with newly diagnosed endometrial cancer undergoing surgery. Lymph node mapping may help in planning surgery to remove endometrial cancer and affected lymph nodes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the detection rate, sensitivity, and negative predictive value of sentinel lymph node (SLN) biopsy in endometrial cancer patients.

SECONDARY OBJECTIVES:

I. To compare different surgical modalities (open procedures, minimally invasive procedures, and single-site technology) and different injectants (isosulfan blue and indocyanine green) for SLN biopsy.

II. To determine total operating room time (from the time the patient enters the room to the time the patient leaves the room) as well as console time (robotic)/operating time for minimally invasive procedures.

OUTLINE:

Patients undergo SLN mapping using isosulfan blue and/or indocyanine green solution injected directly into the cervix. Following SLN identification and biopsy, patients undergo hysterectomy, bilateral salpingo-oophorectomy, and/or complete pelvic lymphadenectomy. Patients expressing SLN positive for metastasis undergo para-aortic lymphadenectomy.

After completion of study treatment, patients are followed up at 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women must have newly diagnosed histologically or cytologically confirmed endometrial cancer
* Women should have received no prior therapy for their disease
* Women who are planning to undergo hysterectomy, bilateral salpingo-oophorectomy, and pelvic lymphadenectomy for the management of their endometrial cancer
* Women must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Women who are receiving any other investigational agents
* Women with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to isosulfan blue or indocyanine green or other agents used in this study
* Women with hypersensitivity to phenylmethane compounds, or a history of allergic reaction to iodides
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women with a history of prior loop electrosurgical excision procedure (LEEP) or cone procedures performed on their cervix
* Women with a history of lymphedema, lymphoma, or lymphatic hyperplasia (Castleman disease)
* Women with a history of a prior malignancy
* Women may also be excluded at the discretion of their surgeon if he or she feels that the patient is not an appropriate candidate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Michener, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Started | 58
Completed | 46
Not Completed | 12
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 7

BASELINE CHARACTERISTICS:
Population: Evaluable participants who completed study
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1
  30-39 years | 0
  40-49 years | 4
  50-59 years | 7
  60-69 years | 21
  70-79 years | 12
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Sentential Lymph Node (SLN) Biopsy
Description: Sensitivity estimated as the proportion of true positives among participants with lymph node metastases. Sensitivity Calculation= the number of patients with a positive SLN over those patients with a positive SLN plus those patients with a false negative lymph node.
Time Frame: Up to 4 weeks
Population: Participants with with lymph node metastases
Measure: Number; unit: percent
Groups:
- Diagnostic (SLN Mapping, Biopsy, Surgery): Participants undergo SLN mapping using isosulfan blue and/or indocyanine green solution injected directly into the cervix. Following SLN identification and biopsy, patients undergo hysterectomy, bilateral salpingo-oophorectomy, and/or complete pelvic lymphadenectomy. Patients expressing SLN positive for metastasis undergo para-aortic lymphadenectomy.
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 13
percent | 100

2. Primary Outcome: Number of Participants in Whom a SLN is Detected
Description: Detection Rate as defined by number of participants in whom a SLN is detected
Time Frame: Up to 4 weeks
Population: Participants who completed study
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
Participants | 44

3. Primary Outcome: Percent of Hemipelvises Identified With SLN
Description: Detection rate, as defined by percent of hemipelvises identified with SLN
Time Frame: Up to 4 weeks
Population: Participants who completed study
Measure: Number; unit: Percent of Hemipelvises
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
Percent of Hemipelvises | 81.5

4. Primary Outcome: Number of Participants With Sentinel Nodes Per Side of Pelvis
Description: Detection rate, as defined as number of participants with a sentinel node found per side of pelvis
Time Frame: Up to 4 weeks
Population: Participants who completed study
Measure: Number; unit: participants
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
participants
  Right side of pelvis | 39
  Left side of pelvis | 36

5. Primary Outcome: False Negative Rate as Defined as Proportion of Participants With False Negative Detection
Description: False negative rate = 1-sensitivity or the number of patients with a false negative SLN over the number of patients with a positive SLN plus those with a false negative lymph node
Time Frame: Up to 4 weeks
Population: Participants who completed study
Measure: Number; unit: Proportion of participants
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
Proportion of participants | 0

6. Primary Outcome: Percent of True Positive SLN Identified With Surgical Modalities (Open Procedures, Minimally Invasive Procedures, and Single-site Technology)
Description: The percent of true positive SLN identified with surgical modalities using pairwise comparisons for each surgical modality. Comparisons will be performed using two sample tests of proportions based on a normal approximation.
Time Frame: Up to 4 weeks
Population: Participants who completed study
Measure: Number; unit: percentage of true positive SNLs
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
percentage of true positive SNLs
  Laparoscopy | 83.3
  Robot | 86.4
  Single port | 79.0

7. Secondary Outcome: Percent of True Positive SLNs Using Isosulfan Blue and Indocyanine Green Solution
Description: Percent of true positive SLN identified will be compared between injectants utilized using a two sample test of proportions based on a normal approximation. Comparisons will be performed using two sample tests of proportions based on a normal approximation.
Time Frame: Up to 4 weeks
Population: Participants who completed study
Measure: Number; unit: Percentage of true positive SLNs
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
Percentage of true positive SLNs
  indocyanine green | 86.54
  Blue dye | 75

8. Secondary Outcome: Total Operating Room Time in Minutes
Description: Total operating room time will be estimated as a mean with 95% confidence interval if the data have an approximately normal distribution. Otherwise, the median and a bootstrapped 95% confidence interval for the median will be reported. Similar summaries will be provided for the console time (robotic)/ operating time.
Time Frame: From the time the patient enters the room to the time the patient leaves the room, assessed up to 4 weeks
Population: Participants who completed study
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
Number analyzed (Participants) | 46
minutes | 158.5 [138.91 to 178.09]

ADVERSE EVENTS:
Time Frame: Up to 30 days from last treatment dose
Arm/Group | Diagnostic (SLN Mapping, Biopsy, Surgery)
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 1/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (SLN Mapping, Biopsy, Surgery) (N=58)
New onset atrial fibrillation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-08-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT01939028/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT01939028/ICF_001.pdf